CLINICAL TRIAL: NCT02609659
Title: An Open-Label, Multicenter Study to Evaluate the Efficacy and Safety of Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir With Low-Dose Ribavirin QD in Subjects With Genotype 1a Chronic Hepatitis C Virus Infection (GEODE II)
Brief Title: Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir With Low-Dose Ribavirin QD in Subjects With Genotype 1a Chronic Hepatitis C Virus Infection
Acronym: GEODE II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M15-582
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Results first posted 2017-10-18 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2017-09

CONDITIONS: Hepatitis C Virus (HCV)
Keywords: Chronic Hepatitis C Infection
MeSH Terms: conditions — Hepatitis C | interventions — ombitasvir; dasabuvir; Viekira Pak; paritaprevir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 3-DAA + RBV 600 mg (Experimental): 3-DAA (ombitasvir/paritaprevir/ritonavir [25 mg/150 mg/100 mg once daily] and dasabuvir [250 mg twice daily]) plus RBV (ribavirin [600 mg once daily]) for 12 weeks.
  Interventions: Drug: ombitasvir/paritaprevir/ritonavir and dasabuvir; Drug: ribavirin

INTERVENTIONS:
Drug: ombitasvir/paritaprevir/ritonavir and dasabuvir — Tablet; ombitasvir coformulated with paritaprevir and ritonavir, dasabuvir tablet
  Other Names: Viekira Pak; paritaprevir also known as ABT-450; ombitasvir also known as ABT-267; dasabuvir also known as ABT-333
Drug: ribavirin — Tablet

SUMMARY:
This study seeks to assess the safety and efficacy of treatment with ombitasvir/paritaprevir/ritonavir and dasabuvir with low-dose ribavirin in non-cirrhotic, genotype 1a (GT1a) hepatitis C virus infected participants who are treatment-naïve or treatment-experienced with Interferon (IFN) or Pegylated Interferon (pegIFN) with or without Ribavirin (RBV).

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C virus (HCV) infection
* Non-cirrhotic subjects
* Screening laboratory results showing HCV Genotype 1a (HCV GT1a) infection
* HCV treatment-naïve or if treated previously, only with interferon (IFN) or pegylated interferon (pegINF) with or without ribavirin (RBV)

Exclusion Criteria:

* Pregnant or breastfeeding women
* Positive for hepatitis B surface antigen (HBsAg) or anti-human immunodeficiency virus antibody (HIV Ab)
* HCV genotype of any subtype other than GT1a or unable to subtype
* Prior or current use of any investigational or commercially available anti-HCV agents other than IFN, pegIFN or RBV. Subjects with previous participation in trials of investigational direct-acting antiviral agents (DAAs) may be enrolled if they can produce documentation that they received only placebo.
* Current enrollment in another interventional clinical study or receipt of any investigational product within 6 weeks prior to study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-10-28 (Actual); Primary Completion 2016-10-07 (Actual); Study Completion 2016-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc, Study Director — AbbVie

REFERENCES:
- [Result] Poordad F, Sedghi S, Pockros PJ, Ravendhran N, Reindollar R, Lucey MR, Epstein M, Bank L, Bernstein D, Trinh R, Krishnan P, Polepally AR, Unnebrink K, Martinez M, Nelson DR. Efficacy and safety of ombitasvir/paritaprevir/ritonavir and dasabuvir with low-dose ribavirin in patients with chronic hepatitis C virus genotype 1a infection without cirrhosis. J Viral Hepat. 2019 Aug;26(8):1027-1030. doi: 10.1111/jvh.13109. Epub 2019 May 6. PMID 30980576
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 3-DAA + RBV 600 mg
Started | 105
Completed | 97
Not Completed | 8
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 6
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | 3-DAA + RBV 600 mg
Number analyzed (Participants) | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (13.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 50

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12)
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification [<LLOQ]) 12 weeks after the last dose of study drug. The primary efficacy endpoint was noninferiority of the percentage of participants who achieved SVR12 in participants in the treatment arm 3-DAA + RBV 600 mg) for 12 weeks compared with the historical control rate for subjects treated with 3-DAA + weight-based RBV for 12 weeks.
Time Frame: 12 weeks after the last actual dose of study drug
Population: Intent-to-treat population: all participants who received at least 1 dose of study drug; participants with missing data after flanking imputation were counted as nonresponders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3-DAA + RBV 600 mg
Number analyzed (Participants) | 105
percentage of participants | 89.5 [83.7 to 95.4]
Statistical Analysis 1: Comparison: 3-DAA + RBV 600 mg; Test type: Non-Inferiority — The noninferiority of the rate of sustained virologic response at 12 weeks after treatment for the 3-DAA + RBV 600 mg treatment group as compared with the historical rate for 3-DAA + weight-based RBV was analyzed; the lower confidence bound of the 2-sided 95% confidence interval (95% CI) for the percentage of participants with sustained virologic response at 12 weeks after treatment must exceed 92% to achieve noninferiority; percentage of participants = 89.5, 95% CI 2-sided [83.7 to 95.4]

2. Primary Outcome: Percentage of Participants With Hemoglobin < 10 g/dL During Treatment
Description: The percentage of participants with hemoglobin <10 g/dL during treatment is provided.
Time Frame: up to 12 weeks
Population: All participants who received at least 1 dose of study drug (ITT population) with at least one post-baseline hemoglobin value through the final treatment value.
Measure: Number; unit: percentage of participants
Arm/Group | 3-DAA + RBV 600 mg
Number analyzed (Participants) | 104
percentage of participants | 0

3. Primary Outcome: Mean Change in Hemoglobin Values From Baseline to End of Treatment
Description: The mean change in hemoglobin (g/L) from baseline to each study visit and to the final treatment visit (up to 12 weeks) is provided.
Time Frame: Baseline (Day 1) to Weeks 2, 4, 8, and 12, and the Final Treatment Visit (up to 12 weeks)
Population: All participants who received at least 1 dose of study drug (ITT population) with a hemoglobin value at baseline and at given timepoint.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | 3-DAA + RBV 600 mg
Number analyzed (Participants) | 104
g/L
  Week 2: number analyzed (Participants) | 102
  Week 2 | -6.4 (8.17)
  Week 4: number analyzed (Participants) | 103
  Week 4 | -8.9 (9.37)
  Week 8: number analyzed (Participants) | 99
  Week 8 | -11.2 (9.85)
  Week 12: number analyzed (Participants) | 89
  Week 12 | -12.4 (10.06)
  Final Treatment Visit | -12.1 (9.90)

4. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as confirmed HCV RNA ≥ LLOQ after HCV RNA < LLOQ during treatment; confirmed increase of > 1 log(subscript)10(subscript) IU/mL above the lowest value post-baseline in HCV RNA during treatment; or all on-treatment values of HCV RNA ≥ LLOQ with at least 6 weeks of treatment.
Time Frame: Up to 12 weeks
Population: All participants who received at least 1 dose of study drug (ITT population).
Measure: Number; unit: percentage of participants
Arm/Group | 3-DAA + RBV 600 mg
Number analyzed (Participants) | 105
percentage of participants | 1.0

5. Secondary Outcome: Percentage of Participants With Post-treatment Relapse
Description: Post-treatment relapse was defined as confirmed HCV RNA ≥ LLOQ between the end of treatment and 12 weeks after the last dose of study drug, excluding reinfection, among participants who completed treatment with HCV RNA levels < LLOQ at the end of treatment.
Time Frame: From the end of treatment through 12 weeks after the last dose of study drug
Population: All participants who received at least 1 dose of study drug, completed treatment, and had HCV RNA <LLOQ at the final treatment visit.
Measure: Number; unit: percentage of participants
Arm/Group | 3-DAA + RBV 600 mg
Number analyzed (Participants) | 97
percentage of participants | 4.1

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from first dose of study drug until 30 days after the last dose of study drug (up to 16 weeks).
Description: TEAEs and TESAEs are defined as any adverse event or serious adverse event that begins or worsens in severity after initiation of study drug until 30 days after the last dose of study drug.
Arm/Group | 3-DAA + RBV 600 mg
Serious Adverse Events (participants affected / at risk) | 3/105
Other Adverse Events (participants affected / at risk) | 53/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 3-DAA + RBV 600 mg (N=105)
CYCLIC VOMITING SYNDROME (Gastrointestinal disorders) | 1
BIPOLAR I DISORDER (Psychiatric disorders) | 1
PSYCHOTIC DISORDER (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 3-DAA + RBV 600 mg (N=105)
CONSTIPATION (Gastrointestinal disorders) | 6
DIARRHOEA (Gastrointestinal disorders) | 9
NAUSEA (Gastrointestinal disorders) | 11
FATIGUE (General disorders) | 29
INFLUENZA (Infections and infestations) | 6
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6
HEADACHE (Nervous system disorders) | 14
ANXIETY (Psychiatric disorders) | 7
INSOMNIA (Psychiatric disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.